CLINICAL TRIAL: NCT01561885
Title: A Pragmatic Randomized Controlled Trial of Patient-Centered Integrated Clinical Pathways Based Versus Usual Care in an Academic Center: National Guard Health Affairs Western Region Experience
Brief Title: Collaborative Healthcare Professionals Approach in Monitoring of Patient Centered Outcomes Through Pathways
Acronym: CHAMP-Path
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Majed Aljeraisy (Other)
Responsible Party: Sponsor-Investigator, Majed Aljeraisy, Research Office Head, King Abdullah International Medical Research Center
Organization: King Abdullah International Medical Research Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RC 10/134/J
Record Dates: First submitted 2012-03-18; First posted 2012-03-23 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Heart Failure; Community Acquired Pneumonia; Venous Thromboembolism; Acute Kidney Injury; Asthma
Keywords: Clinical Pathways; Length of Stay; Patient-Centered Care; Pragmatic Randomized Controlled Trial
MeSH Terms: conditions — Heart Failure; Community-Acquired Pneumonia; Venous Thromboembolism; Acute Kidney Injury; Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients on Pathway Care (Active Comparator)
  Interventions: Other: Pathway-Based Care
- Patients on Usual Care (No Intervention)

INTERVENTIONS:
Other: Pathway-Based Care — Patients who are randomly allocated to Pathway Care will be treated by the Pathway Clinical Teaching Unit as well as other collaborative healthcare professionals (pharmacists, nurses, health educators, nutritionists, and social workers). The Pathway Care physicians will have access to the Clinical Care Plan on the QuadraMed, which is a detailed, organized, day-to-day treatment plan that includes pre-set orders and medications. Physicians for the patients on Usual Care will not have access to this information, and the collaborative healthcare will only be provided upon consultation.
  Arms: Patients on Pathway Care

SUMMARY:
The aim of this study is to determine if by providing a collaborative, integrated pathway-based healthcare compared to the usual healthcare, whether or not this would be superior in reducing the length of hospital stay across five high frequency /high risk medical diagnoses: Acute Venous Thromboembolism, Acute Kidney Injury, Community Acquired Pneumonia, Adult Left Ventricular Heart Failure, and Asthma.

DETAILED DESCRIPTION:
This study is a pragmatic randomized controlled trial. To date, there is a scarcity of randomized controlled trials looking at pathway-based, patient-centered healthcare versus usual care in several high-risk or high volume diagnoses that account for the vast majority of hospitalizations in medical settings.

In this study, the pathway care intervention is a collaborative effort that involves healthcare professionals from multiple departments, including pharmacists, health educators, nurses, social workers, nutritionists, and quality management.

For patients allocated to the usual care, these healthcare professionals will deliver standardized care when consulted. For pathway care patients, this collaborative healthcare will be default.

ELIGIBILITY:
1. Inclusion Criteria (Overall Criteria):

   * One principle diagnosis
   * Hemodynamic Stability
2. Inclusion Criteria (Specific to each Diagnosis):

   Acute Venous Thromboembolism:
   * New onset / in-patient

   Acute Kidney Injury:
   * Patients with increased serum creatinine of more than 50% from baseline

   Community Acquired Pneumonia:
   * Age limit

   Adult Left Ventricular Heart Failure:
   * Age limit

   Asthma
   * Acute exacerbation of Asthma
3. Exclusion Criteria (Overall Criteria):

   * Intensive Care Unit (ICU) patients
   * Pregnancy
4. Exclusion Criteria (Specific to each Diagnosis):

Acute Venous Thromboembolism:

* Hemodynamic instability (Systolic Blood Pressure (SBP) less than 90 mmHg or massive Pulmonary Embolism (PE)
* PE patients with an sPESI Score ≥ 1

Acute Kidney Injury:

* Critical care patients (ICU, Coronary Care Unit, burn units)
* Stage 4 and 5 chronic kidney diseases
* Kidney allograft recipients
* Obstructive uropathy
* Glomerulonephritis
* Interstitial nephritis

Community Acquired Pneumonia:

* Intensive Care Unit (ICU) patients
* Pregnancy

Adult Left Ventricular Heart Failure:

* All non-cardiogenic pulmonary edema
* Patients requiring Inotropic agents

Asthma

* Patients with Chronic Obstructive Pulmonary Disease (COPD) and Bronchiectasis
* Severe Asthma (Peak Expiratory Flow Rate (PEFR) less than 40 percent)

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2012-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Decrease in length of hospital stay by two days | During hospitalization period of 7 to 10 days

SECONDARY OUTCOMES:
30-Day Rehospitalization | After discharge up to 30 days
  To determine the effect of the pathway-based care versus usual care on 30-day rehospitalization rates for the same diagnosis
Determinants of the Length of Stay | Upon admission until discharge
Pathway Care Specific Clinical Outcomes | Upon admission until discharge
  For pathway care, there are specific targeted outcomes that ought to be met.

CONTACTS AND LOCATIONS:
Overall Officials: Mujtaba Quadri, MD, Principal Investigator — National Guard Health Affairs; Sherine Esmail, PharmD, Principal Investigator — National Guard Health Affairs; Saliman Karsou, MD, Principal Investigator — National Guard Health Affairs; Abdulhameed Gasim, MD, Principal Investigator — National Guard Health Affairs; Zeyad Zahrani, MD, Principal Investigator — National Guard Health Affairs; Majed Al Jeraisy, PharmD, Principal Investigator — King Abdullah International Medical Research Center
Locations (1):
- King Khalid National Guard Hospital, Jeddah, Mecca Region, Saudi Arabia